CLINICAL TRIAL: NCT00969163
Title: A Pilot Study to Investigate Biomarkers of Skin Androgenization Following Short-Term Testosterone Administration in Healthy Postmenopausal Women
Brief Title: A Study to Investigate Biomarkers of Skin Androgenization Following Testosterone Administration (0000-015)(COMPLETED).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-015; MK0000-015; 2009_654
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Skin Androgenization
Keywords: Biomarkers of Skin Androgenization
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): 2.5 mg testosterone gel
  Interventions: Drug: testosterone gel
- 2 (Experimental): 300 ug testosterone gel
  Interventions: Drug: testosterone gel
- 3 (Placebo Comparator): placebo gel
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: testosterone gel — 300 ug or 2.5 mg transdermal testosterone gel daily for 6 weeks
  Other Names: AndroGel
  Arms: 1; 2
Drug: Comparator: placebo — transdermal placebo gel for 6 weeks
  Arms: 3

SUMMARY:
Postmenopausal women will receive testosterone gel or matching placebo gel daily. Sebum excretion rates will be measured before and after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 3 years postmenopausal
* Subject is in good general health
* Subject is willing to avoid excess alcohol or strenuous physical activity during the study

Exclusion Criteria:

* Subject has donated a unit of blood or has taken an investigational drug in another clinical trial in the last 4 weeks
* Subject is a regular user of any illicit drugs
* Subject drinks excessive amounts of coffee, tea or cola
* Subject has used an estrogen or progestogens hormone replacement therapy in the past 6 months
* Subject has a history of cancer
* Subject has acne

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2005-04 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
serum free testosterone concentrations following multiple doses of AndroGel | 6 weeks

SECONDARY OUTCOMES:
mean percent change from baseline in sebum excretion | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC